CLINICAL TRIAL: NCT02138448
Title: Implementing Personal Health Records to Promote Evidence-Based Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM15307; 1R01CA168795-01A1 (NIH)
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Health Promotion
Keywords: Cancer Screenings; Health Information Technology; Patient Health Record; Preventive Services
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention practices (Experimental): Intervention practices will implement an interactive preventive health record in addition to their standard personal health record functionality.
  Interventions: Behavioral: Interactive Preventive Health Record
- Control practices (No Intervention): Control practices will continue to field their existing personal health record

INTERVENTIONS:
Behavioral: Interactive Preventive Health Record — The interactive preventive healthcare record (IPHR) is a patient-centered application that links patients to their clinician's record, explains information in lay language, displays tailored recommendations and educational resources, and makes preventive care actionable.
  Other Names: MyPreventiveCare
  Arms: Intervention practices

SUMMARY:
Cancer screening can improve the length and quality of life, yet the average American receives only half of recommended services. Patient-centered personal health records with higher levels of functionality, combined with practice redesign to make use of these functions, can help patients obtain recommended cancer screening tests by linking them to their doctor's records, explaining information in lay language, displaying tailored recommendations and educational resources, providing logistical support and tools to stimulate action, and generating reminders. This project will measure whether making these resources available to primary care practices and patients promotes shared decision-making and increases the delivery of cancer screening compared to existing information systems.

DETAILED DESCRIPTION:
We developed a theory-driven interactive Patient Health Record (PHR) that uses higher functionality to more deeply engage patients in health promotion. The model defines five levels of PHR functionality: (1) collecting patient information, (2) integrating with electronic health records (EHRs), (3) translating information into lay language, (4) providing individualized, guideline-based clinical recommendations, and (5) facilitating patient action. We hypothesize that implementing PHRs with these higher levels of functionality will inform and activate patients in ways that simpler PHRs cannot achieve and will increase uptake of preventive services. In Phase 1, we will randomize 46 practices from three practice-based research networks in eight states to implement a PHR with advanced versus simpler functionality. Control practices will use their existing PHR. Intervention practices will upgrade their PHR to feature an interactive preventive health record (IPHR) that we have previously developed and tested. Intervention practices will locally tailor the IPHR content and learn how to integrate new functions into practice. Phase 1 will feature an implementation assessment in intervention practices, based on the RE-AIM model, to measure Reach (creation of IPHR accounts by patients), Adoption (practice decision to use the IPHR), Implementation (consistency, fidelity, barriers, and facilitators of use), and Maintenance (sustained use). The randomized comparison of intervention and control practices will measure the incremental effect of the IPHR on shared decision-making and receipt of cancer screening tests compared to traditional PHRs (Effectiveness). Data sources will include the EHR/PHR/IPHR databases, patient and practice surveys, recruitment field notes, practice learning collaborative transcripts, practice diaries, and patient phone interviews. This study will inform future efforts to use patient-centered information technology to promote cancer prevention and the feasibility of national dissemination.

ELIGIBILITY:
Inclusion Criteria:

1. Practices in a practice based research network participating in our study that have an existing patient health record
2. Patients that attend our study practices

Exclusion Criteria:

Practices without a patient health record

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Percent of patients who are up-to-date with recommended cancer screening tests in intervention versus control practices. | 1 year
  The percent of eligible patients who are up-to-date with all indicated cancer screenings (all-or-none measure).

SECONDARY OUTCOMES:
Shared decision-making outcomes (knowledge, communication, decisional conflict, and decision control) reported by patients in intervention versus control practices | 1 year
  To assess shared decision making a composite score based on the following measures will be calculated.
  * Knowledge gained will be measured by using the IPHR, we will use questions from NCI's Health Information National Trends Survey (HINTS).
  * To assess whether the IPHR helps patients weigh values regarding risks and benefits 2 measures will be used: (a) process (patient-clinician communication) and (b) patient perception (decisional conflict).
    1. Communication will be measured by using questions from AHRQ's Consumer Assessment of HealthCare Providers and Systems (CAHPS) survey.
    2. O'Connor's low literacy decisional conflict scale will be used to measure decisional conflict.
  * To assess whether the IPHR fosters decision-making engagement at the desired level, Degner's locus of control metric will be used.
To assess whether cancer screening rates differ for disadvantaged patients, defined as minorities and Medicaid beneficiaries. | 1 year
  The difference in delivery of preventive services (Effectiveness) will be calculated for disadvantaged patients and the general population, using a two-level mixed-effects logistic regression for the all-or-none, composite, and individual screening tests.
To assess whether shared decision-making differ for disadvantaged patients, defined as minorities and Medicaid beneficiaries. | 1 year
  To assess shared decision making a composite score based on the following measures will be calculated.
  * Knowledge gained will be measured by using the IPHR, we will use questions from NCI's Health Information National Trends Survey (HINTS).
  * To assess whether the IPHR helps patients weigh values regarding risks and benefits 2 measures will be used: (a) process (patient-clinician communication) and (b) patient perception (decisional conflict).
    1. Communication will be measured by using questions from AHRQ's Consumer Assessment of HealthCare Providers and Systems (CAHPS) survey.
    2. O'Connor's low literacy decisional conflict scale will be used to measure decisional conflict.
  * To assess whether the IPHR fosters decision-making engagement at the desired level, Degner's locus of control metric will be used.
  These scores will be calculated for disadvantaged patients (minorities and Medicaid patients) and the general population that use the IPHR, then compared.
To assess whether perceptions of the technology differ for disadvantaged patients, defined as minorities and Medicaid beneficiaries. | 1 year
  Post-implementation patient phone interviews will be conducted then analyzed using grounded-theory approach to understand disadvantaged patients' perceptions of and experience with the IPHR. These results will be compared to the phone interviews done with patients from the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander H Krist, MD, MPH, Principal Investigator — Virginia Commonwalth University
Locations (3):
- United States (3):
  - University of New Mexico-RIOS Net, Albuquerque, New Mexico
  - OCHIN, Portland, Oregon
  - Virginia Commonwalth University, Richmond, Virginia

REFERENCES:
- [Background] Krist AH, Peele E, Woolf SH, Rothemich SF, Loomis JF, Longo DR, Kuzel AJ. Designing a patient-centered personal health record to promote preventive care. BMC Med Inform Decis Mak. 2011 Nov 24;11:73. doi: 10.1186/1472-6947-11-73. PMID 22115059
- [Background] Krist AH, Woolf SH. A vision for patient-centered health information systems. JAMA. 2011 Jan 19;305(3):300-1. doi: 10.1001/jama.2010.2011. No abstract available. PMID 21245186
- [Background] Kerns JW, Krist AH, Longo DR, Kuzel AJ, Woolf SH. How patients want to engage with their personal health record: a qualitative study. BMJ Open. 2013 Jul 30;3(7):e002931. doi: 10.1136/bmjopen-2013-002931. PMID 23901027
- [Background] Krist AH, Woolf SH, Rothemich SF, Johnson RE, Peele JE, Cunningham TD, Longo DR, Bello GA, Matzke GR. Interactive preventive health record to enhance delivery of recommended care: a randomized trial. Ann Fam Med. 2012 Jul-Aug;10(4):312-9. doi: 10.1370/afm.1383. PMID 22778119
- [Background] Krist AH, Aycock RA, Etz RS, Devoe JE, Sabo RT, Williams R, Stein KL, Iwamoto G, Puro J, Deshazo J, Kashiri PL, Arkind J, Romney C, Kano M, Nelson C, Longo DR, Wolver S, Woolf SH. MyPreventiveCare: implementation and dissemination of an interactive preventive health record in three practice-based research networks serving disadvantaged patients--a randomized cluster trial. Implement Sci. 2014 Dec 11;9:181. doi: 10.1186/s13012-014-0181-1. PMID 25500097
- See also: An Interactive Preventive Care Record: A handbook for implementing patient centered personal health records to promote prevention. — http://healthit.ahrq.gov/sites/default/files/docs/page/PreventiveCareHandbook_062912comp.pdf

DOCUMENTS (1):
  • Informed Consent Form: Focus group consent (2014-01-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT02138448/ICF_000.pdf